CLINICAL TRIAL: NCT00635830
Title: An Open-Label, Single-Dose, Safety and Tolerability Study of Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine in Chinese Female Subjects Aged 9 to 26 Years
Brief Title: An Open-Label, Single Dose Safety Study of Quadrivalent HPV Vaccine in Chinese Female Subjects (V501-035)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V501-035; 2008_003
Record Dates: First submitted 2008-03-03; First posted 2008-03-14 (Estimated); Results first posted 2009-08-20 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

ARMS (1):
- 1 (Experimental): Open Label
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — HPV 6,11,16,18 VLP, 0.5 mL 1 dose injection.
  Other Names: V501

SUMMARY:
To prove that quadrivalent HPV (types 6, 11, 16, 18) L1 virus-like particle (VLP) vaccine is generally safe and well tolerated in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Subject Is Female, Between The Ages Of 9 Years And 0 Days And 26 Years And 364 Days On The Day Of Enrollment
* Subject (Or, For Minor Subjects, Parent/Legal Guardian And Subject) Fully Understands Study Procedures, Alternative Treatments Available, The Risks Involved With The Study, And Voluntarily Agrees To Participate By Giving Written Informed Consent
* Subject Is Able To Read, Understand, And Complete The Vaccination Report Card

Exclusion Criteria:

* Subject Is, At The Time Of Signing Informed Consent, A User Of Recreational Or Illicit Drugs Or Has Had A Recent History (Within The Last Year) Of Drug Or Alcohol Abuse Or Dependence. Alcohol Abusers Are Defined As Those Who Drink Despite Recurrent Social, Interpersonal, And/Or Legal Problems As A Result Of Alcohol Use
* Subject Has A History Of Severe Allergic Reaction (E.G., Swelling Of The Mouth And Throat, Difficulty Breathing, Hypotension Or Shock) That Required Medical Intervention
* Subject Has Known Allergy To Any Vaccine Component, Including Aluminum, Yeast, Or Benzonase (Nuclease, Nycomed [Used To Remove Residual Nucleic Acids From This And Other Vaccines])

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- 18 to 26 Years of Age Group: 18 to 26 years of age group was enrolled to evaluate safety firstly.
  Subjects in this group received one 0.5-ml intramuscular injection of Quadrivalent HPV L1 VLP vaccine.
- 9 to 17 Years of Age Group: 9 to 17 years of age group was enrolled after the Ethics Review Committee approval of the older group safety data.
  Subjects in this group received one 0.5-ml intramuscular injection of Quadrivalent HPV L1 VLP vaccine.
Period: Overall Study
Arm/Group | 18 to 26 Years of Age Group | 9 to 17 Years of Age Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 18 to 26 Years of Age Group | 9 to 17 Years of Age Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.64 (2.39) | 13.82 (9.6) | 18.73 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Body Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 36.64 (0.35) | 36.35 (0.24) | 36.49 (0.33)
Pulse [Mean (Standard Deviation); unit: Beats per minute (BPM)] | 71.75 (4.17) | 65.40 (2.68) | 68.58 (4.72)

OUTCOME MEASURES:

1. Primary Outcome: Measure Serious Adverse Experiences, Systemic Adverse Experiences Occurring Within 14 Days After Vaccination, and Injection-site Complaints Occurring Day 1 Through Day 5 After Vaccination
Description: All adverse experiences were collected from the time the consent form was signed through 14 days following the vaccination. All subjects were requested to record injection-site adverse experiences and monitor temperature daily on the Vaccination Report Card for Day 1 thereafter for 4 additional calendar days, and record all systemic adverse experiences that occur during the 14-day period after injection
Time Frame: For serious adverse experiences and systemic adverse experiences: 14 days follow-up after one dose of vaccination; For injection-site adverse experiences: 5 days follow-up after one dose of vaccination
Measure: Number; unit: Participants
Arm/Group | 18 to 26 Years of Age Group | 9 to 17 Years of Age Group
Number analyzed (Participants) | 20 | 20
Participants
  Serious Adverse Experiences | 0 | 0
  Systemic Adverse Experiences | 7 | 10
  Injection-Site Complaints | 4 | 7

ADVERSE EVENTS:
Arm/Group | 18 to 26 Years of Age Group | 9 to 17 Years of Age Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 10 | 11
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | 18 to 26 Years of Age Group | 9 to 17 Years of Age Group
Injection site painness (General disorders) | 4/20 (4) | 7/20 (7)
Headache (Nervous system disorders) | 0/20 (0) | 3/20 (3)
Conjunctivitis (Eye disorders) | 1/20 (1) | 0/20 (0)
Nausea (Gastrointestinal disorders) | 0/20 (0) | 1/20 (1)
Abdominal pain (Gastrointestinal disorders) | 1/20 (1) | 1/20 (1)
Vomiting (Gastrointestinal disorders) | 0/20 (0) | 1/20 (1)
Gastritis (Gastrointestinal disorders) | 1/20 (1) | 0/20 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 0/20 (0) | 3/20 (3)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0/20 (0) | 2/20 (2)
Menstrual disorder (Reproductive system and breast disorders) | 1/20 (1) | 0/20 (0)
Allergic reaction (General disorders) | 0/20 (0) | 1/20 (1)
Fever (General disorders) | 3/20 (3) | 3/20 (3)
Muscle pain (General disorders) | 0/20 (0) | 3/20 (3)
Fatigue (General disorders) | 1/20 (1) | 2/20 (2)
Hypodynamia (General disorders) | 1/20 (1) | 2/20 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.